CLINICAL TRIAL: NCT07338825
Title: Prevalence of Functional Ankle Instability Among Professional Egyptian Players: a Cross-sectional Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Sherif Maher Mohamed, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/006046
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ankle Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the prevalence of functional ankle instability among professional Egyptian soccer players

ELIGIBILITY:
Inclusion Criteria:

* 1. Three Hundred Soccer players from both genders aged between 8-35 years old including junior teams (8-12 years old), Youth (13-20 years old) and Senior teams (21,>21 years old).

  2. Players have BMI 18-25 (kg/m²). 3. Players are registered in the Egyptian Soccer Association

Exclusion Criteria:

* 1- Systematic pathology that affects balance, reflexes, or muscle strength 2- Lower limb fractures in the 2 years preceding the study 3- Surgery on one of the ankles 4- Structural malalignments 5- Plantar Fasciitis

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Professional Egyptian soccer players
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of functional ankle instability among professional Egyptian soccer players | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt